CLINICAL TRIAL: NCT02695264
Title: Prospective Evaluation of Non-invasive Intracranial Pressure (ICP) Monitoring in Pediatric Patients Undergoing Invasive ICP Monitoring
Brief Title: Non-invasive Intracranial Pressure (ICP) Monitoring in Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical Trial Agreement not executed
Sponsor: HeadSense Medical (Industry)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HS-028
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Intracranial Hypertension
Keywords: intracranial pressure; intracranial hypertension; severe traumatic brain injury
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): ICP readings will be recorded from both the invasive and HeadSense non-invasive ICP monitor for an aggregate of 30 minutes. During the recording sessions, a webcam will take periodic snapshots of the ICP monitor and/or bedside monitor picturing the ICP values and other clinical parameters that are displayed on screen, with a focus on blood pressure and heart rate (HR). Recording sessions will be done until an aggregate of at least 30 minutes of data are collected, depending on the patient's clinical condition. Recording sessions may be repeated over several days until the 30 minute target is reached.
  Interventions: Device: HS-1000 recording

INTERVENTIONS:
Device: HS-1000 recording

SUMMARY:
The purpose of this study is to prospectively evaluate the accuracy and safety of non-invasive intracranial pressure (ICP) measurements using the HeadSense-1000 (HS-1000) device compared to the current invasive external ventricular device (EVD) or parenchymal (bolt) monitoring devices in the pediatric population.

DETAILED DESCRIPTION:
The HS-1000 is an innovative non-invasive intracranial pressure (ICP) monitoring device that employs advanced acoustic signal analysis to derive ICP on a continuous basis. The first version of the device was clinically validated in trials in Italy, India, and Armenia. Overall, more than 10,000 ICP measurements were collected from both patients and healthy subjects. The device is currently undergoing FDA validation in an adult cohort across eight sites in the United States.

This will be a pilot study conducted at Akron Children's Hospital. A maximum of 40 patients with severe traumatic brain injury (TBI) or neurological conditions requiring ICP monitoring will be studied over 2 years. All patients treated with either surgical ICP monitor (external ventricular drain [EVD] or subarachnoid manometer [Bolt]) are eligible for study enrollment. The HS-1000 device will be deployed as soon as possible after surgical ICP monitor placement to record and collect data in parallel with the surgical device.

To assess the accuracy and safety of the HS-1000 device as an alternative to the invasive ICP procedure, the investigators will compare ICP readings obtained by the HS-1000 monitoring system to measurements recorded by the surgical device during 15-30 minute recording sessions.

ICP readings will be recorded from both the invasive and HeadSense non-invasive ICP monitor for an aggregate of 30 minutes. During the recording sessions, a webcam will take periodic snapshots of the ICP monitor and/or bedside monitor picturing the ICP values and other clinical parameters that are displayed on screen, with a focus on blood pressure and heart rate (HR). Recording sessions will be done until an aggregate of at least 30 minutes of data are collected, depending on the patient's clinical condition. Recording sessions may be repeated over several days until the 30 minute target is reached.

The HeadSense headset is removed between recordings. Recording should be done only in case the patient's clinical condition allows it (i.e. patient is in supine position and does not require any clinical intervention or treatment at the time of the recording). In case the patient requires some clinical intervention the recording will be stopped and will be resumed only after the intervention is done and the patient's clinical condition allows resuming of the recording.

Lastly, the investigators will also place a commercial sound meter in the participant's room to collect baseline data on exposure to ambient noise within the Pediatric Intensive Care Unit (PICU) treatment environment. This data will facilitate a device-vs-ambient sound comparison, a component of the device safety profile.

Study patient demographics will be collected to include patient medical record number, age, gender, diagnosis, medical information, and the patient's clinical course pertinent to the ICP monitoring until the attending physician determines invasive ICP measurement is no longer necessary. Additional demographic, diagnostic parameters, severity of illness calculations, and procedures will be obtained from the Virtual Pediatric Systems (VPS, LLC) Pediatric Intensive Care Unit clinical outcomes database. The patient will be followed for 48 hours post ICU discharge for any adverse events.

The diagnosis of head trauma or other medical conditions indicating a need for ICP monitoring, the decision to place an intraventricular catheter and the duration of ICP monitoring are at the discretion of the patient's clinical care team and independent of this study. With the exception of simultaneous use of the non-invasive acoustical HS-1000 monitoring system and ambient noise level measurements within the patient's room, all other patient care, including clinical evaluations and treatments, is independent of this study. No HS-1000 data will be displayed and will not be used in clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Males and females <= 18 years old admitted to the PICU whose treatment includes a surgical ICP monitor.
* Subject or legal authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
* Subject or legal authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

* Subject with an invasive ICP monitor placed Ten (10) days or before the date of recording for EVD monitor OR Five (5) days or before the date of recording for Bolt monitor
* Subjects with more than one invasive ICP monitor in place at the time of recording
* Ear disease/ear trauma
* Subjects with severe head trauma in which the location and/or severity of the skull fracture(s), i.e. frank skull fracture or major joint dislocations with parenchyma exposed to room pressure, may jeopardize HeadSense monitoring procedure [Post-craniotomy patients with intact dura and accurate ICP values from the invasive EVD are eligible.]
* Severe TBI that jeopardizes HS-1000 monitoring procedure
* Cerebral spinal fluid (CSF) otorrhea
* Allergy/Hypersensitivity to test materials
* Pregnant or breast feeding
* Current enrollment (or within 30 days) in another investigational device or drug study, OR receiving an investigational agent
* Any condition that jeopardizes study participation (abnormal clinical/lab finding)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ICP recordings from the HS-1000 device compared to those from the invasive ICP monitor | 5 days of bolt insertion or 10 days of EVD insertion

SECONDARY OUTCOMES:
Safety of the HS-1000 as determined by number of reported device-related adverse events | Up to 48hours after last recording

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Forbes, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No